CLINICAL TRIAL: NCT04074668
Title: CROCODILE Study: Control of Renal Oxygen Consumption, Mitochondrial Dysfunction, and Insulin Resistance
Brief Title: Control of Renal Oxygen Consumption, Mitochondrial Dysfunction, and Insulin Resistance
Acronym: CROCODILE
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 19-1282
Record Dates: First submitted 2019-08-06; First posted 2019-08-30 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Kidney Disease; Type 1 Diabetes; Diabetes; Diabetes Mellitus; Diabetes Complications; Diabetic Nephropathies; Type1diabetes; Diabetes, Autoimmune; Autoimmune Diabetes; Juvenile Diabetes; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 1; Diabetes Mellitus; Diabetes Complications | interventions — p-Aminohippuric Acid; Iohexol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — During the study, blood and urine samples will be collected for assessment of kidney function and kidney injury markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 1 Diabetes: All participants will undergo DXA scan, magnetic resonance imaging (MRI) studies of the kidneys, PET/CT using 11-C acetate to measure renal oxygen consumption, hyperinsulinemic-euglycemic clamp to quantify insulin sensitivity, and renal clearance testing using iohexol and para-aminohippurate (PAH) to quantify glomerular filtration rate (GFR) and effective renal plasma flow (ERPF).
  Interventions: Drug: Aminohippurate Sodium Inj 20%; Drug: Iohexol Inj 300 milligrams/milliliter (mg/ml); Radiation: PET/CT Scan; Procedure: Renal Biopsy
- Healthy Controls: All participants will undergo DXA scan, magnetic resonance imaging (MRI) studies of the kidneys, PET/CT using 11-C acetate to measure renal oxygen consumption, hyperinsulinemic-euglycemic clamp to quantify insulin sensitivity, and renal clearance testing using iohexol and para-aminohippurate (PAH) to quantify glomerular filtration rate (GFR) and effective renal plasma flow (ERPF).
  Interventions: Drug: Aminohippurate Sodium Inj 20%; Drug: Iohexol Inj 300 milligrams/milliliter (mg/ml); Radiation: PET/CT Scan; Procedure: Renal Biopsy

INTERVENTIONS:
Drug: Aminohippurate Sodium Inj 20% — Diagnostic aid/agent used to measure effective renal plasma flow (ERPF)
  Other Names: Sodium 4-amino hippurate (PAH) inj 20% 2 grams (g)/10 milliliters (mL); Para-aminohippurate; Aminohippuric acid
Drug: Iohexol Inj 300 milligrams/milliliter (mg/ml) — Diagnostic aid/agent used to measure glomerular filtration rate (GFR)
  Other Names: omnipaque 300
Radiation: PET/CT Scan — Imaging used to visualize the kidneys and quantify renal metabolic activity
Procedure: Renal Biopsy — Minimally invasive outpatient procedure to obtain renal tissue after ultrasound visualization.

SUMMARY:
Type 1 diabetes (T1D) is a complex metabolic disorder with many pathophysiological disturbances including insulin resistance (IR) and mitochondrial dysfunction which are causally related to the development of diabetic kidney disease (DKD) and which contribute to reduced life expectancy. Renal hypoxia, stemming from a potential metabolic mismatch between increased renal energy expenditure and impaired substrate utilization, is increasingly proposed as a unifying early pathway in the development of DKD. By examining the interplay between factors responsible for increased renal adenosine triphosphate (ATP) consumption and decreased ATP generation in young adults with and without T1D, this study hopes to identify novel therapeutic targets to impede the development of DKD in future trials.

The investigators propose to address the specific aims in a cross-sectional study with 30 adults with T1D and 20 controls without a diagnosis of diabetes. For this protocol, participants will complete a one day study visit at Children's Hospital Colorado. Patients will undergo a Dual-energy X-Ray Absorptiometry (DXA) scan to assess body composition, renal Magnetic Resonance Imaging (MRI) to quantify renal oxygenation and perfusion, and a Positron Emission Tomography/Computed Tomography (PET/CT) scan to quantify renal O2 consumption. After the PET and MRI, participants will undergo a hyperinsulinemic-euglycemic clamp to quantify insulin sensitivity. Glomerular Filtration Rate (GFR) and Effective Renal Plasma Flow (ERPF) will be measured by iohexol and PAH clearances during the hyperinsulinemic-euglycemic clamp. To further investigate the mechanisms of renal damage in T1D, two optional procedures are included in the study: 1) kidney biopsy procedure and 2) induction of induced pluripotent stem cells (iPSCs) to assess morphometrics and genetic expression of renal tissue.

ELIGIBILITY:
Inclusion Criteria -- Type 1 Diabetes:

* Antibody positive Type 1 Diabetes with duration > 5 years
* BMI between 18.5 and 30 kg/m2
* Weight < 350 lbs
* HbA1c < 11%
* Hemoglobin >= 12 g/dl

Exclusion Criteria -- Type 1 Diabetes:

* Recent diagnosis (within 3 months) of Diabetic Ketoacidosis (DKA)
* Severe illness
* Pregnancy, nursing
* Anemia
* Allergy to shellfish or iodine
* Claustrophobia or implantable metal devices (MRI contraindications)
* High blood pressure (greater than 130/80 mm Hg)
* Elevated Urine Albumin-to-Creatinine Ratio (UACR) (>30 mg/g) or estimated Glomerular Filtration Rate (eGFR) <90 ml/min/1.73 m2
* Taking ACE inhibitors (ACEis), Angiotensin receptor blockers (ARBs), diuretics, Sodium Glucose Transporter (SGLT) 1/2 blockers

Inclusion Criteria -- Healthy Controls:

* No diagnosis of Type 1 or Type 2 Diabetes
* BMI between 18.5 and 30 kg/m2
* Weight < 350 lbs
* HbA1c < 11%
* Hemoglobin >= 12 g/dl

Exclusion Criteria -- Healthy Controls:

* Severe illness
* Pregnancy, nursing
* Anemia
* Allergy to shellfish or iodine
* Claustrophobia or implantable metal devices (MRI contraindications)
* High blood pressure (greater than 130/80 mm Hg)
* Elevated UACR (>30 mg/g) or eGFR <90 ml/min/1.73 m2
* Taking ACE inhibitors (ACEis), Angiotensin receptor blockers (ARBs), diuretics, SGLT 1/2 blockers

Additional exclusion criteria for participants undergoing optional kidney biopsy:

* Evidence of bleeding disorder or complications from bleeding
* Use of aspirin, NSAIDS or other blood thinner that cannot be safely stopped for a sufficient time period before and after the biopsy so as to add no additional risk of bleeding
* Blood urea nitrogen (BUN) > 80 gm/dL
* INR > 1.4
* PTT > 35 seconds
* Hemoglobin (Hgb) < 10 mg/dL
* Platelet count < 100,000 / µL
* Uncontrolled or difficult to control hypertension (> 150/90 mmHg at the day of biopsy)
* eGFR < 40 mL/min/1.73m2
* Single kidney (either by history, documented by prior imaging or ultrasound performed prior to the biopsy)
* > 2 cm discrepancy between left and right kidney sizes based on largest longitudinal diameter determined by ultrasound performed prior to the biopsy.
* Kidney size: One or both kidneys < 9 cm
* Hydronephrosis or other important renal ultrasound findings such as significant stone disease
* Any evidence of a current urinary tract infection as indicated on day of biopsy
* Clinical evidence of non-diabetic renal disease
* Positive urine pregnancy test or pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We propose to address the specific aims of this study in a cross-sectional project with 30 adults with T1D and 20 controls (50% female, ages 18-30 yr).
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Renal Oxygenation | 30 minutes
  Blood oxygen level dependent (BOLD) MRI
Renal Perfusion | 30 minutes
  Arterial Spin Labeling (ASL) MRI
Renal Oxygen Consumption | 30 minutes
  11-C Acetate PET/CT
Insulin Sensitivity | 4.5 hours
  Hyperinsulinemic-Euglycemic Clamp
Mitochondrial Function | 5 minutes
  Blood draw for mitochondrial DNA copy number
Mitochondrial Function | 5 minutes
  Blood draw for untargeted metabolite assessment of the tricyclic acid (TCA) cycle
Mitochondrial Function | 5 minutes
  Blood draw for targeted assessment and quantification of glucose oxidation using an established metabolite panel
Mitochondrial Function | 5 minutes
  Blood draw for untargeted metabolite assessment of Free Fatty Acid (FFA) oxidation

SECONDARY OUTCOMES:
Glomerular Filtration Rate (GFR) | 3 hours
  Iohexol Clearance Study
Effective Renal Plasma Flow (ERPF) | 2.5 hours
  PAH Clearance Study
Renin-Angiotensin-Aldosterone-System Activity | 5 minutes
  Blood draw for Plasma Renin levels
Renin-Angiotensin-Aldosterone-System Activity | 5 minutes
  Blood draw for Angiotensin II levels
Renin-Angiotensin-Aldosterone-System Activity | 5 minutes
  Blood draw for Copeptin levels
Kidney Injury Biomarkers | 5 minutes
  Blood draw for Tyrosine Lysine Leucine-40 (YKL-40) levels
Kidney Injury Biomarkers | 5 minutes
  Blood draw for Neutrophil gelatinase-associated lipocalin (NGAL) levels
Kidney Injury Biomarkers | 5 minutes
  Blood draw for Kidney Injury Marker 1 (KIM-1) levels
Kidney Injury Biomarkers | 5 minutes
  Blood draw for Interleukin-18 (IL-18) levels
Kidney Injury Biomarkers | 5 minutes
  Blood draw for Tumor Necrosis Factor Receptor 1/2 (TNF-R 1/2) levels

OTHER OUTCOMES:
Podocyte numerical density and number per glomerulus | 4 hours
  Measured by light microscopy from tissue obtained by renal biopsy
Foot process width of glomeruli | 4 hours
  Measured by electron microscopy from tissue obtained by renal biopsy
Detachment and endothelial fenestration of glomeruli | 4 hours
  Measured by electron microscopy from tissue obtained by renal biopsy
Podocyte volume of glomeruli | 4 hours
  Measured by electron microscopy from tissue obtained by renal biopsy
Number and identity of RNA in kidney cells | 4 hours
  Measured from tissue obtained by renal biopsy
Epigenetic profiling | 4 hours
  Measured from tissue obtained by renal biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi YJ, Richard G, Zhang G, Hodgin JB, Demeke DS, Yang Y, Schaub JA, Tamayo IM, Gurung BK, Naik AS, Nair V, Birznieks C, MacDonald A, Narongkiatikhun P, Gross S, Driscoll L, Flynn M, Tommerdahl K, Nadeau KJ, Shah VN, Vigers T, Snell-Bergeon JK, Kendrick J, van Raalte DH, Li LP, Prasad P, Ladd P, Chin BB, Cherney DZ, McCown PJ, Alakwaa F, Otto EA, Brosius FC, Saulnier PJ, Puelles VG, Goodrich JA, Street K, Venkatachalam MA, Ruiz A, de Boer IH, Nelson RG, Pyle L, Blondin DP, Sharma K, Kretzler M, Bjornstad P. Attenuated kidney oxidative metabolism in young adults with type 1 diabetes. J Clin Invest. 2024 Oct 22;134(24):e183984. doi: 10.1172/JCI183984. PMID 39436695
- [Derived] Bjornstad P, Richard G, Choi YJ, Nowak KL, Steele C, Chonchol MB, Nadeau KJ, Vigers T, Pyle L, Tommerdahl K, van Raalte DH, Hilkin A, Driscoll L, Birznieks C, Hopp K, Wang W, Edelstein C, Nelson RG, Gregory AV, Kline TL, Blondin D, Gitomer B. Kidney Energetics and Cyst Burden in Autosomal Dominant Polycystic Kidney Disease: A Pilot Study. Am J Kidney Dis. 2024 Sep;84(3):286-297.e1. doi: 10.1053/j.ajkd.2024.02.016. Epub 2024 Apr 15. PMID 38621633